CLINICAL TRIAL: NCT01874873
Title: Phase 2 Study of Anlotinib in Advanced Medullary Thyroid Carcinoma
Brief Title: A Phase II Study of Anlotinib in MTC Patients
Acronym: ALTN/MTC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-01-IIA
Record Dates: First submitted 2013-05-30; First posted 2013-06-11 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Tumor
MeSH Terms: conditions — Neoplasms | interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anlotinib (Experimental)
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib
  Other Names: ALTN

SUMMARY:
Anlotibib (ALTN) is a kind of innovative medicines approved by State Food and Drug Administration（SFDA） which was researched by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd. ALTN is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR2 and VEGFR3. It has the obvious resistance to new angiogenesis. The trial is to explore ALTN for the effectiveness of advanced medullary thyroid carcinoma and security.

ELIGIBILITY:
Inclusion Criteria:

* 1.late medullary thyroid carcinoma; 2.18-70years, ECOG:0-2,Expected survival period >3 months; 3.Calcitonic≥500pg/ml, thyroid function normal; 4.HB≥100g/L,ANC(Absolute Neutrophil Count) ≥1.5×109/L；PLT

  * 80×109/L ,BIL/Cr in normal range,ALT/AST(aspartate aminotransferase )≤1.5*ULN(for hepatic metastases,ALT/AST(aspartate aminotransferase )≤5*ULN) ;TG≤ 3.0mmol/L，cholesterol≤7.75mmol/L; LVEF
  * LLN. 5.Username contraceptive during the study and after 6 months; 6.Volunteer.

Exclusion Criteria:

* 1.Received vascular endothelial growth inhibitor type of targeted therapy; 2.Subject was diagnosed with The second cancer; 3.Participated in other clinical trials in four weeks; 4.Received in other radiotherapy or chemotherapy treatment in four weeks; 5.With AE> 1; 6.Has influence of oral drugs; 7.Brain metastases, spinal cord compression, cancerous meningitis, or the brain/soft meningeal disease patient; 8.Any serious or failed to control the disease 9.Artery/venous thrombotic; 10.Coagulant function abnormality; 11.Arteriovenous thrombosis event; 12.History of psychiatric drugs abuse or a mental disorder; 13.Immunodeficiency history; 14.Concomitant diseases.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
enhanced CT scan | each 42 days up to 48 months

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | each 21 days up to up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Jinwan Wang, doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Pingzhang Tang, doctor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (10):
- China (10):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The first hospital affiliated to fujian medical university, Fuzhou, Fujian
  - Gansu Province Tumor Hospital, Lanzhou, Gansu
  - Sun Yat-Sen University Cancer Center, Guozhou, Guangdong
  - Harbin medical university affiliated tumor hospital, Harbin, Heilongjiang
  - Jiangsu province tumor hospital, Nanjing, Jiangsu
  - Liaoning Province Tumor Hospital, Shenyang, Liaoning
  - Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality